CLINICAL TRIAL: NCT06085170
Title: Voice Analysis in Women With Polycystic Ovary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Wafaa Helmy Abdelhakeem, Principal Investigator, Minia University
Other Study IDs: voice character in PCO
Record Dates: First submitted 2023-08-20; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Voice Change
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Group I (women with PCOs on ultrasound)
  Interventions: Diagnostic Test: Acoustic Analysis by MDVP
- Group II: group II(Group II will be women rated to have a normal voice as assessed using Auditory-Perceptual Evaluation of Voice, these women have a regular menstrual cycles and no PCOS on ultrasound)
  Interventions: Diagnostic Test: Acoustic Analysis by MDVP

INTERVENTIONS:
Diagnostic Test: Acoustic Analysis by MDVP — Acoustic measurements: Acoustic analysis using Multidimensional voice program software (MDVP) will be carried out with the sustained /a/vowel for 9 seconds, for measuring frequency, jitter, shimmer and harmonic to noise ratio of the voice

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder affecting up to one in five reproductive-aged women.

It is associated with clinical and/or biochemical hyperandrogenism, oligomenorrhea, and polycystic appearance of ovaries in ultrasonography. Voice changes have been traditionally recognized as a feature of PCOS for years. However, voice analyses of patients with PCOS are limited. The human larynx is a highly hormone-sensitive target with the presence of hormonal receptors within the vocal folds, and vocal changes occur in relation to the fluctuations in the sex hormones. During the reproductive years and throughout the menstrual cycle, vocal changes have been reported in almost one-third of nonprofessional voice users.The aim of this work is to evaluate the voice characteristics among women with PCOS

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder affecting up to one in five reproductive-aged women.

It is associated with clinical and/or biochemical hyperandrogenism, oligomenorrhea, and polycystic appearance of ovaries in ultrasonography. Voice changes have been traditionally recognized as a feature of PCOS for years. However, voice analyses of patients with PCOS are limited. The human larynx is a highly hormone-sensitive target with the presence of hormonal receptors within the vocal folds, and vocal changes occur in relation to the fluctuations in the sex hormones. During the reproductive years and throughout the menstrual cycle, vocal changes have been reported in almost one-third of nonprofessional voice users. Hyperandrogenism is a landmark in the diagnosis of PCOS, and androgen-related voice changes in women have been recognized.The aim of this work is to evaluate the voice characteristics among women with PCOS The study will include 50 women with and without PCOS. They will divided into 2 groups. Group I will comprise of the 25 women in the clinical group diagnosed with PCOS on ultrasound, while Group II will comprise of 25 typical women as controls Patients will be selected from Obstetric gynecological clinics of El Minna University Hospital .This study is approved by the ethics committee in the Faculty of medicine, Minna university hospital, and concents will be obtained from subjects.

Methods

1. History taking.
2. Abdominal ultrasonography
3. voice sample by recording (in sustained vowel |a| )
4. Auditory Perceptual Assessment (APA)
5. Arabic voice handicap index (VHI): For measurement of the voice severity with the Arabic version of VHI
6. laryngoscopic examination Patients will taken to a room with a tower on which the 8.5 mm 70 rigid laryngoscopic (KARL STORZ - endoscope) (Tele pack X LED).
7. Acoustic analysis: The voice sample will be subjected to computerized acoustic analysis using Multidimensional voice program software(MDVP).

The results will be presented in tables and charts.Statistical analysis:Parametric and non-parametric tests included in statistical package for social science version 19 .The level of significance for this study is at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Group I participants:

  * women with polycystic ovaries on ultrasound.
* Group II will be:

  * women have a regular menstrual cycles and no PCOS on ultrasound

Exclusion Criteria:

* Women with hypersensitive gag reflex,
* alcohol consumption,
* Smoking,
* reflux symptoms and vocal abuse will be excluded in both groups.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 50 women with and without PCOS They will divided into 2 groups. Group I will comprise of the 25 women in the clinical group diagnosed with PCOS on ultrasound, while Group II will comprise of 25 typical women as controls
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
frequency | baseline
  frequency in hertz
jitter | baseline
  jitter in percentage%
shimmer | baseline
  shimmer in decibel
Harmonic to noise ratio | baseline
  Harmonic to noise ratio in decibel

CONTACTS AND LOCATIONS:
Overall Officials: Hany G Eissawy, MD, Study Chair — Minia University

REFERENCES:
- [Background] Hannoun A, Zreik T, Husseini ST, Mahfoud L, Sibai A, Hamdan AL. Vocal changes in patients with polycystic ovary syndrome. J Voice. 2011 Jul;25(4):501-4. doi: 10.1016/j.jvoice.2009.12.005. Epub 2010 May 26. PMID 20537860
- [Result] Aydin K, Akbulut S, Demir MG, Demir S, Ozderya A, Temizkan S, Sargin M. Voice characteristics associated with polycystic ovary syndrome. Laryngoscope. 2016 Sep;126(9):2067-72. doi: 10.1002/lary.25818. Epub 2015 Dec 23. PMID 26700739